CLINICAL TRIAL: NCT01078831
Title: Intrabronchial Airway Pressures in Intubated Patients During Bronchoscopy Under Volume Controlled (VC) and Pressure Controlled (PC) Ventilation
Brief Title: Intrabronchial Airway Pressures in Intubated Patients During Bronchoscopy
Status: Completed | Type: Observational
Sponsor: Oslo University Hospital (Other)
Responsible Party: Fredrik Borchsenius, MD, Head of Department for Pulmonary Medicine, Oslo University Hospital
Other Study IDs: REK-HO Ref 191-01055, 03052001
Record Dates: First submitted 2010-03-01; First posted 2010-03-02 (Estimated); Last update posted 2010-11-11 (Estimated); Status verified 2010-11

CONDITIONS: Acute Respiratory Distress Syndrome; Acute Lung Injury (ALI)
MeSH Terms: conditions — Respiratory Distress Syndrome; Acute Lung Injury | interventions — Bronchoscopy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Arterial blood gases
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- ARDS / ALI patients
  Interventions: Other: Bronchoscopy

INTERVENTIONS:
Other: Bronchoscopy — Airway pressures, ventilation changes and blood gas changes are recorded in a group of intubated patients on mechanical ventilation before and after bronchoscope insertion. The registration is done immediately before a therapeutic/diagnostic bronchoscopy requested by a staff physician not involved n the study.

SUMMARY:
The purpose of this study is to examine changes in ventilation and airway pressures during conventional bronchoscopy of intubated patients.

DETAILED DESCRIPTION:
Mechanically ventilated patients often need bronchoscopy as a diagnostic procedure or for visually directed elimination of secretions. Partial endotracheal tube occlusion by the bronchoscope increases airflow resistance. Inhibition of inspiratory flow may be compensated for by augmented inspiratory pressure. Reduced expiratory flow however, cannot be compensated for by most ventilators and could lead to higher airway - and intrathoracic pressures that are not detected by pressure transducers in the ventilator tubing. In this study we compare changes in ventilation, airway pressures, ventilator pressures and blood gases during bronchoscopy of intubated patients in both volume controlled and pressure controlled ventilation. Our hypothesis are that 1) increased resistance in the tube during bronchoscopy leads to high intrabronchial airway pressures when the ventilator is in volume controlled mode, and 2) when the ventilator is in pressure controlled mode, increased resistance in the tube during bronchoscopy leads to reduced Tidal Volume and moderately increased paCO2.

ELIGIBILITY:
Inclusion Criteria:

* ARDS/ALI patients on mechanical ventilation
* endotracheal tube size 7-9mm
* age > 18 years
* therapeutic or diagnostic bronchoscopy requested by staff physician

Exclusion Criteria:

* SpO2 < 90%
* unstable BP
* pneumothorax
* acute cardiovascular disease
* cerebrovascular or other condition that requires stable BP and saturation

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: ARDS/ALI patients on mechanical ventilation where a therapeutic or diagnostic bronchoscopy has been requested by the staff physician.
Sampling Method: Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2002-03; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
Changes in ventilation, airway pressures and blood gases after bronchoscope insertion. | 2 minutes after bronchoscope insertion/ mode change
  paO2, paCO2 (kPa), airway and ventilator pressures (cmH2O)

CONTACTS AND LOCATIONS:
Overall Officials: Helge Opdahl, MD, PhD, Study Director — Oslo University Hospital - Ulleval, Norway; Ole H Skjønsberg, MD, PhD, Study Director — Ullevaal University Hospital; Fredrik Borchsenius, MD, Study Director — Ullevaal University Hospital
Locations (1):
- Oslo University Hospital - Ulleval, Oslo, Oslo County, Norway